CLINICAL TRIAL: NCT06380855
Title: Flexible Colonoscope Assisted Hybrid Transanal Total Mesorectal Resection (taTME)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Flexible Colonoscope Assisted Hybrid Transanal Total Mesorectal Resection (taTME), Sun Yat-sen University
Other Study IDs: GIHSYSU-34
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Flexible colonoscope assisted taTME group: Flexible colonoscope assisted hybrid transanal total mesorectal resection (taTME) group
  Interventions: Procedure: Flexible colonoscope assisted hybrid transanal total mesorectal resection

INTERVENTIONS:
Procedure: Flexible colonoscope assisted hybrid transanal total mesorectal resection — Endoscopic pursestring suture (EPSS) was performed at the distance from 1cm to the inferior edge of the tumor by a double-channel flexible colonoscope. An endoloop was inserted through one channel. Meanwhile, the endoclips was inserted through the other channel one by one to fix the endoloop around the rectal wall. And then the endoloop was tightened slowly. After completing the routine lavage lumen, a full-thickness, circumferential dissection was performed by flexible colonoscope following taTME surgical principle until it converged with the laparoscopy group.

SUMMARY:
The investigators propose to use flexible endoscopy combined with transanal total mesorectal resection to further reduce anal injury.

DETAILED DESCRIPTION:
Endoscopic technique has become an indispensable part of Natural orifice transluminal endoscopic surgery (NOTES). However, the upper gastrointestinal tract is easy to cause severe leakage complications, which mainly limits the application of endoscopy in rectum. Herein, investigators propose purse suture closing distal rectum and full-layer incision of the rectal wall using flexible endoscopic from anal to assist in hybrid transanal total mesorectal resection (taTME).Further reduce the damage of anus caused by taTME.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old
2. Confirmed rectal adenocarcinoma cancer pathologically
3. tumor location ≦ 12 cm from the anal margin
4. Willing and able to provide written informed consent for participation in this study

Exclusion Criteria:

1. distant metastasis before surgery
2. more than one colorectal tumor at diagnosis
3. familial adenomatous polyposis
4. recurrent rectal cancer
5. undergo transanal minimally invasive surgery
6. undergo palliative treatment
7. undergo emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients suitable for transanal endoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-08-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
Success rate of operation | 1 years after the surgery
  Whether it is necessary to switch to other surgical methods

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided